CLINICAL TRIAL: NCT02240160
Title: A Randomised, Open-label, Three-way Crossover Study to Assess the Pharmacokinetics and Safety of Single Doses of Four Sprays of Sativex® in a Range of Oral pH Environments in Healthy Subjects
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: GW Pharmaceuticals Ltd (Industry)
Responsible Party: Sponsor
Organization: GWPharm (Unknown)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: GWCP10116; 2013-004459-19 (EudraCT Number)
Record Dates: First submitted 2014-09-11; First posted 2014-09-15 (Estimated); Last update posted 2021-02-05 (Actual); Status verified 2021-02

CONDITIONS: Healthy Volunteers
Keywords: Sativex; Pharmacokinetics; Oral pH
MeSH Terms: conditions — Marijuana Abuse | interventions — nabiximols

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Sativex: acidic oral pH (Experimental): Four sprays of Sativex taken within two minutes of pH measurement immediately following oral pre-treatment with Coca-Cola (30 mL held in the mouth for 45-60 seconds then spat out, repeated three times).
  Interventions: Drug: Sativex
- Sativex: neutral oral pH (Experimental): Four sprays of Sativex taken within two minutes of pH measurement immediately following oral pre-treatment with tap water (30 mL held in the mouth for 45-60 seconds then spat out, repeated three times).
  Interventions: Drug: Sativex
- Sativex: alkaline oral pH (Experimental): Four sprays of Sativex taken within two minutes of pH measurement immediately following oral pre-treatment with milk of magnesia (30 mL held in the mouth for 45-60 seconds then spat out, repeated three times).
  Interventions: Drug: Sativex

INTERVENTIONS:
Drug: Sativex — Oromucosal spray containing THC (27 mg/mL) and CBD (25 mg/mL) in ethanol:propylene glycol (50:50) excipients, with peppermint oil (0.05%) flavouring. Each 100 μL spray delivers 2.7 mg THC and 2.5 mg CBD.
  Other Names: Nabiximols; THC/CBD spray

SUMMARY:
To evaluate the effect of oral pH on the pharmacokinetics (PK) of a single oromucosal dose of Sativex (four sprays containing 10.8 mg Δ9 tetrahydrocannabinol (THC) and 10 mg cannabidiol (CBD)) by comparing the PK profile of Sativex in healthy subjects.

The primary clinical hypothesis is that there will be an effect of oral pH on the PK of Sativex when administered as a single oromucosal dose (four sprays).

DETAILED DESCRIPTION:
This is a Phase I, randomised, open-label, three-way crossover study to assess the effects of oral pH on the PK of Sativex. Subjects will receive each of the following treatments in a random order across three residential treatment visits:

* Treatment A (acidic oral pH): Sativex (four sprays) after pre-treatment with Coca-Cola;
* Treatment B (neutral oral pH): Sativex (four sprays) after pre-treatment with tap water;
* Treatment C (alkaline oral pH): Sativex (four sprays) after pre-treatment with an oral suspension of magnesium hydroxide (milk of magnesia).

The target pH for each treatment will be determined from the results of a pilot study.

Each dose administration will be separated by at least seven days. Study subjects will participate in a total of five study visits.

ELIGIBILITY:
Inclusion Criteria:

* Subject is willing and able to give informed consent for participation in the study;
* Male and/or female subjects aged 18 to 50 years, inclusive;
* Subject must weigh at least 50.0 kg and have a body mass index (BMI) between 19.0 and 35.0 kg/m2, inclusive;
* Subject must be a non-smoker for at least three months prior to screening and must be willing to abstain from smoking during the study;
* Subject must be in good health as determined by the investigator from medical history, physical and oral examination findings, 12-lead standard ECG findings and clinical laboratory test results (laboratory results outside of the reference range must be documented as acceptable by both the investigator and sponsor);
* Subject is able (in the investigator's opinion) and willing to comply with all study requirements;
* Subject is willing to allow his or her primary care practitioner and consultant, if appropriate, to be notified of participation in the study.

Exclusion Criteria:

* Use of any prescription medications or herbal supplements within 2 weeks prior to Day 1 of the first treatment visit or any over the counter medications or supplements within 72 hours prior to first study medication administration;
* Subject has oral issues/condition likely, in the opinion of the investigator, to affect the assessment of the oromucosal absorption of Sativex;
* Subject is physically dependent on alcohol, has a history of drug or alcohol abuse within the 12 months prior to dose administration or evidence of such abuse as indicated by the laboratory assays conducted during the screening or baseline evaluations;
* Subject has a positive result for the presence of hepatitis B surface antigen (HBsAg), hepatitis C virus antibodies (HCAb) or human immunodeficiency virus (HIV) antibodies;
* Subject is currently using or has used cannabis, cannabinoid-based medications (e.g. Marinol®, Nabilone®, Cannador®) or Acomplia (rimonabant) or taranabant within 30 days of study entry (first treatment visit) and is unwilling to abstain for the duration of the study;
* Subject consumes more than five caffeinated beverages per day (e.g., five cups of tea or coffee or cans of cola) or is unwilling to abstain from consumption of caffeine-containing food and beverages throughout the study period;
* Subject has any known or suspected history or family history of schizophrenia, or other psychotic illness, history of severe personality disorder or other significant psychiatric disorder;
* Subject has any history of epilepsy as evidenced by one or more seizures in the last 12 months;
* Subject has any known or suspected hypersensitivity to cannabinoids or any of the excipients of the investigational medicinal product (IMP), Coca-Cola or antacid medications;
* Subject who has received an IMP within the 12 weeks prior to the screening visit, or who has received the last dose of an IMP greater than three months ago but is on extended follow-up;
* Subject with any other significant disease or disorder which, in the opinion of the investigator, may either put the subject at risk because of participation in the study, may influence the result of the study or the subject's ability to participate in the study;
* Following a physical examination, the subject has any abnormalities that, in the opinion of the investigator would prevent the subject from safe participation in the study;
* Travel outside the country of residence planned during the study;
* Subjects who are vegans or have medical dietary restrictions.
* Subject has a positive urine drug (including THC), cotinine or alcohol result at screening or at Day -1 of first treatment visit; or positive urine drug (excluding THC), cotinine or alcohol result at Day -1 of subsequent treatment visits;
* Female subjects of child bearing potential and male subjects whose partner is of child bearing potential, unless willing to ensure that they or their partner use two effective forms of contraception e.g, oral contraception, double barrier or intra-uterine device (IUD), during the study and for three months thereafter (however a male condom should not be used in conjunction with a female condom);
* Female subject who is pregnant, lactating or planning pregnancy during the course of the study and for three months thereafter;
* Subjects who have donated or lost more than 450 mL of blood in the 60 days prior to screening or are unwilling to abstain from donation of blood during the study;
* Subject has previously been randomised into this study.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 6 (Actual)
Dates: Start 2014-08; Primary Completion 2014-08 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic parameters of THC: Cmax, AUC(0-t), and AUC(0-∞) | 0-24 hours post-dose
  Mean highest observed plasma concentration of the measured concentration-time profile (Cmax), area under the concentration-time curve from administration to the last sampling point (AUC(0-t)), and area under the concentration-time curve extrapolated to infinity (AUC(0-∞)) of THC are presented.
Pharmacokinetic parameters of CBD: Cmax, AUC(0-t), and AUC(0-∞) | 0-24 hours post-dose
  Mean Cmax, AUC(0-t), and AUC(0-∞) of CBD are presented.

SECONDARY OUTCOMES:
Pharmacokinetic parameters of 11-hydroxy-CBD (11-OH-CBD): Cmax, AUC(0-t), and AUC(0-∞) | 0-24 hours post-dose
  Mean Cmax, AUC(0-t), and AUC(0-∞) of 11-OH-CBD are presented.
Pharmacokinetic parameters of 7-hydroxy-CBD (7-OH-CBD): Cmax, AUC(0-t), and AUC(0-∞) | 0-24 hours post-dose
  Mean Cmax, AUC(0-t), and AUC(0-∞) of 7-OH-CBD are presented.
Pharmacokinetic parameters of 6-hydroxy-CBD (6-OH-CBD): Cmax, AUC(0-t), and AUC(0-∞) | 0-24 hours post-dose
  Mean Cmax, AUC(0-t), and AUC(0-∞) of 6-OH-CBD are presented.
Pharmacokinetic parameters of THC: t½ and Tmax | 0-24 hours post-dose
  Mean terminal elimination half-life (t½) and time to maximum plasma concentration (Tmax) of THC are presented.
Pharmacokinetic parameters of 11-OH-CBD: t½ and Tmax | 0-24 hours post-dose
  Mean t½ and Tmax of 11-OH-CBD are presented.
Pharmacokinetic parameters of CBD: t½ and Tmax | 0-24 hours post-dose
  Mean t½ and Tmax of CBD are presented.
Pharmacokinetic parameters of 7-OH-CBD: t½ and Tmax | 0-24 hours post-dose
  Mean t½ and Tmax of 7-OH-CBD are presented.
Pharmacokinetic parameters of 6-OH-CBD: t½ and Tmax | 0-24 hours post-dose
  Mean t½ and Tmax of 6-OH-CBD are presented.
Total body clearance (CL/F) of THC and CBD from plasma | 0-24 hours post-dose
  Mean total body clearance of THC and CBD from plasma is presented.
The incidence of adverse events as measure of subject safety | From screening to follow-up, an expected average of 35 days
  The number of subjects who experienced an adverse event during the study is presented. The time-frame for adverse event reporting was from screening to the follow-up visit.
The number of subjects with a clinically significant change in physical and oral examination results, relative to pre-treatment baseline | From screening to follow-up, an expected average of 35 days
  The number of subjects with a change in physical and oral examination results indicative of an adverse event, relative to the pre-treatment baseline, is presented.
The number of subjects with a clinically significant change in 12-lead electrocardiogram (ECG) results, relative to pre-treatment baseline | From screening to follow-up, an expected average of 35 days
  The number of subjects with a change in ECG results indicative of an adverse event, relative to the pre-treatment baseline, is presented.
The number of subjects with clinically significant changes in laboratory test parameters, relative to pre-treatment baseline | From screening to follow-up, an expected average of 35 days
  The number of subjects with clinically significant changes in serum biochemistry, haematology and urinalysis, relative to the pre-treatment baseline, is presented.
The number of subjects with a clinically significant change in vital signs, relative to pre-treatment baseline | From screening to follow-up, an expected average of 35 days
  The number of subjects with a change in vital signs (systolic blood pressure, diastolic blood pressure, pulse rate) indicative of an adverse event, relative to the pre-treatment baseline, is presented.
The number of subjects with a clinically significant change in body temperature, relative to pre-treatment baseline | From screening to follow-up, an expected average of 35 days
  The number of subjects with a change in body temperature indicative of an adverse event, relative to the pre-treatment baseline, is presented.
The number of subjects with a clinically significant change in body weight, relative to pre-treatment baseline | From screening to follow-up, an expected average of 35 days
  The number of subjects with a change in body weight indicative of an adverse event, relative to the pre-treatment baseline, is presented.

CONTACTS AND LOCATIONS:
Overall Officials: James Ritter, DPhil, FRCP, FMedSci, Principal Investigator — Quintiles Drug Research Unit at Guy's Hospital, Quintiles Ltd, 6 Newcomen Street, London SE1 1YR, United Kingdom